CLINICAL TRIAL: NCT02022566
Title: The Effect of Structured Information and Individually Adapted Exercise on Levels of Physical Activity Measured by Accelerometer in Patients With Knee or Hip Osteoarthritis - an Observational Study With Control Group.
Brief Title: Effect of Structured Info and Adapted Exercise in OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vastra Gotaland Region (Other Government); The Swedish Rheumatism Ass (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 747-08
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis knee; Osteoarthritis hip; Physical activity; accelerometer
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Motor Activity

ARMS (2):
- Supported self-management of osteoarthrits program (Experimental): Treatment with an supported self-management program for osteoarthritis.
  Interventions: Behavioral: A supported self management of osteoarthritis program
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: A supported self management of osteoarthritis program — Three theoretical sessions, each of about 90 minutes, held as group sessions with about 10 participants in each group. After the intervention patients are offered an individual exercise program, and the opportunity to practice this program together with others under supervision of a physical therapist for 6 weeks.
  Arms: Supported self-management of osteoarthrits program

SUMMARY:
Physical activity level is measured at baseline and after 3 and 12 months after structured information and individually adapted exercise for patients with osteoarthritis in hip or knee.

The hypothesis of this study is that a supported self management of osteoarthritis program will increase the level of physical activity in patients with osteoarthritis in hip or knee. The second hypothesis is that patients with osteoarthritis in knee will increase their level of physical activity more than patients with osteoarthritis in hip.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of our most common chronic joint disorders. The World Health Organization (WHO) has estimated that every second woman and every fourth man over the age of 60 suffer some form of OA. OA is most common in hands, knee, hip and back. OA is a rheumatic disorder which affects the whole joint and may start as early as in the age of 30. The main symptoms are pain, stiffness and decreased quality of life.

The primary goals of OA management are to reduce the symptoms. Patient education and exercises are recommended as basic treatment according to national as well as international guidelines.

It is known that the level of physical activity decreases with age and that woman are less physical active than men. A study of healthy women older than 56 years showed that the level of activity decreased by 10 minutes per year, for every five year increase in age. OA is more common in women and is an irreversible disease, which means that the proportion of older women with osteoarthritis is large.

In addition OA is the most common cause of inactivity among the elderly and many fear that activity will further damage the joints. Inactivity is a large risk factor for poor physical and psychological health as well as premature death. Level of physical activity in people with OA has mainly been evaluated by self-assessment questionnaires. People with hip OA are more active than people with knee OA and the correlation between the degree of radiographic changes and physical activity is weak. Only 30% with early OA of the knee in the age group 35-65 years meet the recommendations for physical activity performed at least 30 minutes per day of moderate intensity, five days per week, measured by an accelerometer.

The primary aim of this study is to determine the effects of structured information and individually adapted exercises, delivered as a supported self-management osteoarthritis program, on overall levels of physical activity of moderate and vigorous intensity in patients with hip or knee OA. The secondary aim is to compare the level of physical activity in patients with hip and knee OA.

Supported self-management program for patients with osteoarthritis has been studied before and it's shown that it improves the quality of life, the physical function and decrease pain. No studies have investigated the effect of supported self-management on the level of physical activity.

This is an observational study with control group. Assessments are made at baseline and at 3 and 12 month after the supported self-management course.

The self-management program comprise three theoretical sessions, each of about 90 minutes, led by a physical therapist and held as group sessions with about 10 participants in each group. On the third session an osteoarthritis communicator participates. That is a person with osteoarthritis who communicate the lifestyle changes he/she have done to live a good life with OA. After the theoretical part the patients are offered an individually adapted exercise program, and the opportunity to practice this program together with others under supervision of a physical therapist twice per week for 6 weeks. Patients are also encouraged to find one or two exercises to perform continuously as home exercises. During the program home exercise and other alternatives as changing activity, using walking sticks, pain management ect are introduced in order to maintain the level of physical activity over an extended period of time. The importance of being physically active for a long time is accentuated in all aspects of the patient education. The primary aim of the supported self-management program is to increase the level of physical activity and empower patients to manage their disease, avoid illness and live a good life despite osteoarthritis.

Physical activity is measured with an accelerometer at baseline, 3 month and 12 month. We will also study the correlation between objectivity measured physical activity with physical activity questionnaire (UCLA), quality of life (EQ-5D), pain (VAS 0-100) and comorbidity.

All subjects in our study are also registered in a Swedish national quality register called Better management of patients with osteoarthritis (BOA). Some of the data used in the present study are collected from the register.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old.
2. Patients with clinically verified OA, coming to see a physical therapist for the Supported self-management of osteoarthritis program.

Exclusion Criteria:

1. Other serious disorders causing hip or knee pain (e.g. tumor, rheumatic arthritis, sequel hip fracture).
2. Other symptoms more aggravating than the OA problem (e.g. chronic pain, fibromyalgia, cardio-respiratory dysfunction, spinal condition).
3. Total joint replacement surgery within the past 12 months.
4. Other surgery of knee or hip within the past 3 months.
5. Unable to read and understand Swedish and follow verbal and visual instructions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carina A Thorstensson, Ass prof, Principal Investigator — Göteborg University
Locations (1):
- Skånes universitets sjukhus, Lund, Sweden

REFERENCES:
- [Derived] Jonsson T, Ekvall Hansson E, Thorstensson CA, Eek F, Bergman P, Dahlberg LE. The effect of education and supervised exercise on physical activity, pain, quality of life and self-efficacy - an intervention study with a reference group. BMC Musculoskelet Disord. 2018 Jun 21;19(1):198. doi: 10.1186/s12891-018-2098-3. PMID 30037339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because of a large drop out from the Accelerometer assessment, we recruit more participants
Period: Overall Study
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Started | 227 | 90
Completed | 169 | 49
Not Completed | 58 | 41

BASELINE CHARACTERISTICS:
Population: The intervention group have been a part of a supported self-management of osteoarthritis and the control group were sign to meet a orthopedic doctor because of problems from knee or hip.
Groups:
- Total: Total of all reporting groups
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group | Total
Number analyzed (Participants) | 195 | 69 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 66 (7) | 64 (9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 125 | 40 | 165
  men | 70 | 29 | 99
BMI [Mean (Standard Deviation); unit: kg/m2] | 28 (5) | 28 (5) | 28 (5)
Joint [Count of Participants; unit: Participants]
  knee | 152 | 38 | 190
  hip | 43 | 31 | 74
Education [Count of Participants; unit: Participants]
  elementary school | 47 | 24 | 71
  high school | 78 | 25 | 103
  university | 70 | 20 | 90
Charnley Category (A=unilateral hip-OA, B=bilateral hip-OA, C=multiple joint OA [Count of Participants; unit: Participants]
  A | 55 | 24 | 79
  B | 81 | 23 | 104
  C | 59 | 22 | 81
Sedentary daily minutes [Median (Inter-Quartile Range); unit: minutes] | 562 [523 to 605] | 572 [505 to 599] | 565 [520 to 602]
Low activity daily minutes [Median (Inter-Quartile Range); unit: minutes] | 180 [150 to 214] | 169 [130 to 218] | 178 [145 to 215]
Moderate-vigorous activity daily minutes [Median (Inter-Quartile Range); unit: minutes] | 34 [22 to 52] | 20 [11 to 30] | 30 [19 to 45]
Visual Analogue Scale pain (0 to 100, 0=no pain, 100=worst imaginable pain [Median (Inter-Quartile Range); unit: units on a scale] | 51 [36 to 62] | 60 [50 to 70] | 54 [42 to 64]
EuroQol 5 Dimension index, minimal value -0.594 (worst health), maximal value 1.00 (best health) [Median (Inter-Quartile Range); unit: EQ-5D index] | 0.725 [0.62 to 0.796] | 0.656 [0.159 to 0.727] | 0.692 [0.48 to 0.757]
Arthritis Self-Efficacy Scale-other symptoms, Likert scale 10-100, (10 worst, 100 best) [Median (Inter-Quartile Range); unit: units on a scale (10-100)] | 68 [53 to 80] | 61 [48 to 70] | 66 [51 to 78]
Arthritis Self-Efficacy Scale-pain, Likert scale 10-100, 10 worst, 100 best [Median (Inter-Quartile Range); unit: units on a scale (10-100)] | 60 [46 to 76] | 46 [38 to 62] | 58 [44 to 72]

OUTCOME MEASURES:

1. Primary Outcome: Level of Physical Activity/Sedentary Time
Description: The level of physical activity will be monitored by a GT1M Actigraph which is a small uniaxial accelerometer that measures vertical acceleration and deceleration. Accelerometer output is an activity "count" which is the weighted sum of the number of accelerations measured over a period (e.g. in this case 10 seconds). Participants will be instructed to wear the accelerometer from the morning, and continuously (except for water activities) until going to bed at night, for seven consecutive days. The accelerometer will be attached to a belt to wear around the waist with accelerometer placement on the right hip. The account of minutes in sedentary time will be calculated and the average of minutes in one week will be used.
Time Frame: Baseline, 3 months and 12 months
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 141 | 52
minutes
  baseline | 562 [523 to 605] | 572 [505 to 599]
  3 months | 556 [507 to 602] | 556 [504 to 592]
  12 months | 552 [499 to 598] | NA [NA to NA] — The control group is only measured with baseline and 3 month follow-up
Statistical Analysis 1: Comparison: Supported Self-management of Osteoarthrits Program vs Control Group; Test type: Other; p < 0.05, ANOVA

2. Primary Outcome: Level of Physical Activity/Low Activity
Description: Level of physical activity will be monitored by an accelerometer at baseline and at 3 and 12 months after the supported self-management of osteoarthritis program using an accelerometer. The GT1M Actigraph is a small uniaxial accelerometer that measures vertical acceleration and deceleration. Accelerometer output is an activity "count" which is the weighted sum of the number of accelerations measured over a period (e.g. in this case 10 seconds).
  Participants will be instructed to wear the accelerometer from morning, and continuously (except for water activities) until going to bed at night, for seven consecutive days. The accelerometer will be attached to a belt to wear around the waist with accelerometer placement on the right hip.
Time Frame: baseline, 3 months and12 months
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 141 | 52
minutes
  baseline | 181 [150 to 214] | 169 [130 to 218]
  3 months | 170 [144 to 205] | 169 [118 to 220]
  12 months | 178 [140 to 228] | NA [NA to NA] — The control group was only had 3 month follow-up
Statistical Analysis 1: Comparison: Supported Self-management of Osteoarthrits Program vs Control Group; Test type: Other — Described elsewhere; p < 0.05, ANOVA; Mean Difference (Final Values) = 0.05

3. Primary Outcome: Level of Physical Activity/Moderate-vigorous Activity
Description: as for outcome 2
Time Frame: baseline, 3 month and 12 month
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 141 | 52
minutes
  baseline | 34 [22 to 52] | 20 [11 to 30]
  3 month | 34 [19 to 52] | 21 [10 to 37]
  12 month | 32 [18 to 52] | NA [NA to NA] — The control group only had follow-up at 3 month

4. Secondary Outcome: Health Realted Quality of Life
Description: To evaluate the health-related quality of life the EQ-5D-3L has been used. In this study, we have used the index of EQ-5D-3L with a British tariff. This scale is between (i.e., minimal value -0.594 (worst health), maximal value 1.00 (best health).
Time Frame: baseline, 3 months and 12 months
Measure: Median (Inter-Quartile Range); unit: eq-5d index
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 193 | 69
eq-5d index
  baseline | 0.73 [0.62 to 0.80] | 0.66 [0.16 to 0.73]
  3 months | 0.73 [0.69 to 0.80] | 0.52 [0.09 to 0.73]
  12 months | 0.73 [0.69 to 0.80] | NA [NA to NA] — The control group is only measured at baseline and 3 month follow-up

5. Secondary Outcome: Visual Analog Scale for Pain
Description: Visual Analog Scale for Pain has been used to evaluate pain. This is a scale from 0-100 mm there higher scores indicating higher intensity of pain. We have asked for the average pain the last month.
Time Frame: baseline, 3 months and 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 195 | 69
units on a scale
  baseline | 51 [36 to 62] | 60 [50 to 70]
  3 months | 37 [21 to 54] | 62 [37 to 71]
  12 months | 38 [21 to 57] | NA [NA to NA] — The control group only have 3 month follow-up.

6. Secondary Outcome: Arthritis Self-efficacy Scale/Pain (ASES)
Description: The Arthritis Self-Efficacy Scale (ASES) is a widely used self-report measure of beliefs reflecting confidence in one's capacity to function despite pain and control pain or other symptoms of arthritis. ASES is scored on a 10-point Likert scale ranging from 10 (very uncertain=worst) to 100 (very certain=best).
Time Frame: baseline, 3 months and 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 193 | 69
units on a scale
  baseline | 60 [46 to 76] | 46 [38 to 62]
  3 months | 74 [56 to 86] | 50 [32 to 70]
  12 months | 68 [46 to 84] | NA [NA to NA] — Control group only followed up at 3 month

7. Post Hoc Outcome: Arthritis Self-efficacy Scale/Other Symptoms
Description: as for outcome 6
Time Frame: baseline, 3 months and 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
Number analyzed (Participants) | 193 | 69
units on a scale
  baseline | 68 [53 to 80] | 61 [48 to 70]
  3 months | 76 [61 to 86] | 56 [46 to 81]
  12 months | 71 [55 to 83] | NA [NA to NA] — Control group only followed up at 3 month

ADVERSE EVENTS:
Time Frame: 12 month
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Supported Self-management of Osteoarthrits Program | Control Group
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/195 | 0/69
Other Adverse Events (participants affected / at risk) | 0/195 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes